CLINICAL TRIAL: NCT00385970
Title: A Phase III Trial Comparing UFT+PSK to UFT+LV in Stage IIB, III Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Multicenter Clinical Study Group of Osaka, Colorectal Cancer Treatment Group (Other)
Responsible Party: Principal Investigator, Masataka Ikeda, MD, PhD., Associate Director of Surgery, Osaka National Hospital, Multicenter Clinical Study Group of Osaka, Colorectal Cancer Treatment Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCSGO-CCTG-0501
Record Dates: First submitted 2006-10-08; First posted 2006-10-11 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tegafur; Leucovorin; polysaccharide-K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): UFT+LV Group: The group treated with UFT and LV
  Interventions: Drug: Tegafur-uracil (UFT); Drug: Calcium folinate (LV)
- 2 (Experimental): UFT+PSK Group: The group treated with of UFT and PSK
  Interventions: Drug: Tegafur-uracil (UFT); Drug: Krestin (PSK)

INTERVENTIONS:
Drug: Tegafur-uracil (UFT) — From within 9 weeks after surgery, 300 mg/m2, PO from day 1 to day 28 of each 35 day cycle. Number of Cycles: 5
  Other Names: UFT
Drug: Calcium folinate (LV) — From within 9 weeks after surgery, 75 mg, PO from day 1 to day 28 of each 35 day cycle. Number of Cycles: 5
  Other Names: LV
  Arms: 1
Drug: Krestin (PSK) — From within 9 weeks after surgery to 12 months after surgery, 3 g/day, PO every day
  Other Names: PSK
  Arms: 2

SUMMARY:
To compare the efficacy of tegafur/uracil (UFT) plus folinate calcium (leucovorin: LV) administered orally and UFT plus Krestin (PSK) administered orally enrolling patients with pTNM stage IIB or III colorectal cancer as subjects in a multicenter collaborative randomized open-label comparative controlled study and consequently to determine the usefulness of the above regimens as adjuvant therapy after surgery.

DETAILED DESCRIPTION:
To compare the efficacy of tegafur/uracil (UFT) plus folinate calcium (leucovorin: LV) administered orally and UFT plus Krestin (PSK) administered orally enrolling patients with pTNM stage IIB or III (UICC Sixth version) colorectal cancer/histological curability A (Japanese Classification of Colorectal Carcinoma, Sixth version) as subjects in a multicenter collaborative randomized open-label comparative controlled study and consequently to determine the usefulness of the above regimens as adjuvant therapy after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pTNM stage IIB or III (UICC Sixth version) primary colon cancer/rectal cancer who have undergone surgery of histological curability A (including laparoscopic surgery) (the curability is judged after surgery)
* Patients with primary tumor that directly invades other organs or structures and/or perforates into the visceral peritoneum (T4) or with histologically positive lymph node metastasis (N+) (to be judged after surgery)
* Patients who is between 20 and 80 years old at the time of obtaining informed consent
* Patients with performance status of 0 - 2
* Patients without receiving any cancer treatment such as radiation, chemotherapy, and immunotherapy before surgical operation
* Patients without severe dysfunction of renal, hepatic, or bone marrow function
* Patients without serious complications such as bone marrow suppression, diarrhea, and infections diseases
* Patients who have given consent to participate in this clinical study by himself/herself or his/her family

Exclusion Criteria:

* Patients in whom the bottom of tumor reaches the peritoneal reflection
* Patients with lower rectal cancer (Rb), anal canal (P), or circumanal skin (E)
* Patients who has active multiple cancers or whose disease-free survival is less than 5 years even though the cancers are metachronous (except carcinoma in situ and skin cancers)
* Women who are currently pregnant or wish to be pregnant during this clinical study
* Patients who are judged to be inappropriate to participate in this clinical study by the investigator or subinvestigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2006-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
3-Year recurrence-free survival rate | 3-years after surgery

SECONDARY OUTCOMES:
5-Year survival rate, incidence of adverse events, treatment compliance, QOL, type of metastasis/recurrence, and 3-year and 5-year recurrence-free survival rates and survival rates based on each parameter including colon/rectum, stage, and IAP. | 5-years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Morito Monden, MD, PhD, Study Chair — Multicenter Clinical Study Group of Osaka
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

REFERENCES:
- [Background] Ohwada S, Ikeya T, Yokomori T, Kusaba T, Roppongi T, Takahashi T, Nakamura S, Kakinuma S, Iwazaki S, Ishikawa H, Kawate S, Nakajima T, Morishita Y. Adjuvant immunochemotherapy with oral Tegafur/Uracil plus PSK in patients with stage II or III colorectal cancer: a randomised controlled study. Br J Cancer. 2004 Mar 8;90(5):1003-10. doi: 10.1038/sj.bjc.6601619. PMID 14997197